CLINICAL TRIAL: NCT02938286
Title: Parameters in Fractional Laser Assisted Delivery of Topical Anesthetics: Role of Laser Type and Laser Settings
Brief Title: Fractional Laser Assisted Delivery of Anesthetics III
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Netherlands Institute for Pigment Disorders (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NL53766.018.15
Record Dates: First submitted 2016-10-09; First posted 2016-10-19 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Local Anesthesia of the Skin
Keywords: Fractional laser; Topical anesthesia; Drug delivery; CO2 laser; Er:YAG laser
MeSH Terms: interventions — Carticaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fractional CO2 laser at 5% density (Experimental): This test region will be pretreated with a fractional carbon dioxide laser with a 120 μm spot at 5% density and a pulse energy of 2.5 mJ/microbeam (Fractional CO2 laser, 2.5 mJ, 5% density) in a subject blinded fashion. After pretreament Articaine hydrochloride 40 mg/ml and epinephrine 10 μg/ml solution (AHES) will be applied to this test region. Fifteen minutes after AHES application (incubation time; under occlusion), a pain stimulus will be given at the test region with the Fractional CO2 laser, 50 mJ, 5% density.
  Interventions: Device: Fractional CO2 laser, 2.5 mJ, 5% density; Device: Fractional CO2 laser, 50 mJ, 5% density; Drug: AHES
- Fractional CO2 laser at 15% density (Experimental): This test region will be pretreated with a fractional carbon dioxide laser with a 120 μm spot at 15% density and a pulse energy of 2.5 mJ/microbeam (Fractional CO2 laser, 2.5 mJ, 15% density) in a subject blinded fashion. After pretreament Articaine hydrochloride 40 mg/ml and epinephrine 10 μg/ml solution (AHES) will be applied at this test region. Fifteen minutes after AHES application (incubation time; under occlusion), a pain stimulus will be given at the test region with the Fractional CO2 laser, 50 mJ, 5% density.
  Interventions: Device: Fractional CO2 laser, 2.5 mJ, 15% density; Device: Fractional CO2 laser, 50 mJ, 5% density; Drug: AHES
- Fractional Er:YAG laser at 5% density (Experimental): This test region will be pretreated with a Erbium Yttrium Aluminum Garnet laser with a 225 μm spot at 5% density and a pulse energy of 9 mJ/microbeam (Fractional Er:YAG laser, 9 mJ, 5% density) in a subject blinded fashion. After pretreatment Articaine hydrochloride 40 mg/ml and epinephrine 10 μg/ml solution (AHES) will be applied at this test region. Fifteen minutes after AHES application (incubation time; under occlusion), a pain stimulus will be given at the test region with the Fractional CO2 laser, 50 mJ, 5% density.
  Interventions: Device: Fractional Er:YAG laser, 9 mJ, 5% density; Device: Fractional CO2 laser, 50 mJ, 5% density; Drug: AHES
- Fractional Er:YAG laser at 15% density (Experimental): This test region will be pretreated with a Erbium Yttrium Aluminum Garnet laser with a 225 μm spot at 15% density and a pulse energy of 9 mJ/microbeam (Fractional Er:YAG laser, 9 mJ, 15% density) in a subject blinded fashion. After pretreatment Articaine hydrochloride 40 mg/ml and epinephrine 10 μg/ml solution (AHES) will be applied at this test region. Fifteen minutes after AHES application (incubation time; under occlusion), a pain stimulus will be given at the test region with the Fractional CO2 laser, 50 mJ, 5% density.
  Interventions: Device: Fractional Er:YAG laser, 9 mJ, 15% density; Device: Fractional CO2 laser, 50 mJ, 5% density; Drug: AHES

INTERVENTIONS:
Device: Fractional CO2 laser, 2.5 mJ, 5% density — Pretreatment at 2.5 mJ/microbeam and 5% density. Pain stimulus at 50 mJ/microbeam and 5% density
  Other Names: Fractional carbon dioxide laser; UltraPulse®, DeepFx handpiece; Lumenis Inc.; Ablative fractional laser
  Arms: Fractional CO2 laser at 5% density
Device: Fractional CO2 laser, 2.5 mJ, 15% density — Pretreatment at 2.5 mJ/microbeam and 15% density. Pain stimulus at 50 mJ/microbeam and 5% density
  Other Names: Fractional carbon dioxide laser; UltraPulse®, DeepFx handpiece; Lumenis Inc.; Ablative fractional laser
  Arms: Fractional CO2 laser at 15% density
Device: Fractional Er:YAG laser, 9 mJ, 5% density — Pretreatment at 9 mJ and 5% density.
  Other Names: Fractional Erbium Yttrium Aluminum Garnet laser; P.L.E.A.S.E.® Professional; Pantec Biosolutions; Ablative fractional laser
  Arms: Fractional Er:YAG laser at 5% density
Device: Fractional Er:YAG laser, 9 mJ, 15% density — Pretreatment at 9 mJ and 15% density.
  Other Names: Fractional Erbium Yttrium Aluminum Garnet laser; P.L.E.A.S.E.® Professional; Pantec Biosolutions; Ablative fractional laser
  Arms: Fractional Er:YAG laser at 15% density
Device: Fractional CO2 laser, 50 mJ, 5% density — Pain stimulus at 50 mJ/microbeam and 5% density
  Other Names: Fractional carbon dioxide laser; UltraPulse®, DeepFx handpiece; Lumenis Inc.; Ablative fractional laser
Drug: AHES — Topical application at test region I-IV under occlusion for 15 minutes
  Other Names: Ultracain D-S forte; Articaine hydrochloride 40 mg/ml + epinephrine 10 μg/ml

SUMMARY:
The purpose of this study is to compare the effect of pretreatment with two different ablative laser modalities, a CO2 laser and an Er:YAG laser, and to assess the role of laser density in fractional laser assisted topical anesthesia.

DETAILED DESCRIPTION:
Rationale: In dermatology anesthetics are frequently injected or topically applied to achieve local anesthesia. Injectable anesthetics are effective but uncomfortable during administration, especially for people who are needle phobic. Application of topical anesthesia is painless but time consuming and often only partial aesthesia is achieved due to the barrier function of the stratum corneum. (Manuskiatti, Triwongwaranat et al. 2010) Penetration of local anesthetics could be enhanced by pretreatment of the skin with ablative fractional lasers (AFXL) which locally disrupts the stratum corneum by creating an array of microscopic ablation channels. (Sklar, Burnett et al. 2014) In a previous pilot study, conducted at our institute, we demonstrated that effective anesthesia could be achieved within ten minutes after application of a topical anesthetic on skin pretreated with AFXL at painless settings. (Meesters, Bakker et al. 2015) However, little is still known about the role of the type of fractional laser used (e.g. CO2 or Er:YAG laser), the laser settings, the type of anesthetic and the occlusion time on the efficacy of the anesthesia.

Objective: The objectives of this study are to compare the efficacy of pretreatment with two different ablative laser modalities, a CO2 laser and an Er:YAG laser, and to assess the role of laser density in fractional laser assisted topical anesthesia.

Study design: Prospective, single blinded, randomized, controlled, within subject, pilot study.

Study population: 15 healthy volunteers ≥18 years, who give written informed consent Intervention: In each subject, four test regions on subject's back of 1x1 cm will be randomly allocated to (I) pretreatment with the fractional CO2 laser at 5% density, (II) pretreatment with the fractional CO2 laser at 15% density, (III) pretreatment with the fractional Er:YAG laser at 5% density and (IV) pretreatment with the fractional Er:YAG laser at 15% density. After pretreatment, articaine hydrochloride 40 mg/ml + epinephrine 10 μg/ml 30 solution (AHES) will be applied on the test regions with 15 minutes occlusion time. After 15 minutes a pain stimulus, consisting of a pass with the fractional CO2 laser at 50 mJ and 5% density (scanned area 6x6 mm), will be given at each test region. In addition, a reference pain stimulus with the CO2 laser at the same settings will be given at unanesthetized skin. Subjects will be asked to indicate pain on a visual analogue scale (VAS) from 0-10 (0: no pain; 10: worst imaginable pain) directly after each pain stimulus.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin type I or II
* Age ≥18 years
* Patient is willing and able to give written informed consent

Exclusion Criteria:

* History of keloid or hypertrophic scar formation or complicated wound healing
* Presence of any active skin disease
* Known allergy to local anesthesia
* Pregnancy or lactation
* Incompetency to understand what the procedure involves
* Current complaints of chronic pain or other alterations in pain sensation (e.g. due to diabetes mellitus or lepra)
* Current treatment with systemic analgesics or other medication that can influence pain sensation
* Current treatment with anticoagulants
* Fitzpatrick skin type III-VI
* Excessive sun tan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pain score | After 15 minutes incubation time of the anesthetics
  The main study parameter is pain, as scored on a VAS from 0-10 (0: no pain; 10: worst imaginable pain).

SECONDARY OUTCOMES:
Pain score | Directly after pretreatment.
  The secondary study parameter is pain, as scored on a VAS from 0-10 (0: no pain; 10: worst imaginable pain) directly after pretreatment

CONTACTS AND LOCATIONS:
Overall Officials: Albert Wolkerstorfer, MD, PhD, Principal Investigator — Netherlands Institute for Pigment Disorders, Department of Dermatology, Academic Medical Center, University of Amsterdam; Menno A. De Rie, MD, PhD, Study Director — Department of Dermatology, Academic Medical Center, University of Amsterdam
Locations (1):
- Netherlands Institute for Pigment Disorders, Amsterdam, Netherlands

REFERENCES:
- [Background] Meesters AA, Bakker MM, de Rie MA, Wolkerstorfer A. Fractional CO2 laser assisted delivery of topical anesthetics: A randomized controlled pilot study. Lasers Surg Med. 2016 Feb;48(2):208-11. doi: 10.1002/lsm.22376. Epub 2015 May 29. PMID 26032635
- [Background] Sklar LR, Burnett CT, Waibel JS, Moy RL, Ozog DM. Laser assisted drug delivery: a review of an evolving technology. Lasers Surg Med. 2014 Apr;46(4):249-62. doi: 10.1002/lsm.22227. Epub 2014 Mar 24. PMID 24664987
- [Background] Oni G, Brown SA, Kenkel JM. Can fractional lasers enhance transdermal absorption of topical lidocaine in an in vivo animal model? Lasers Surg Med. 2012 Feb;44(2):168-74. doi: 10.1002/lsm.21130. Epub 2012 Feb 2. PMID 22302761
- [Background] Oni G, Rasko Y, Kenkel J. Topical lidocaine enhanced by laser pretreatment: a safe and effective method of analgesia for facial rejuvenation. Aesthet Surg J. 2013 Aug 1;33(6):854-61. doi: 10.1177/1090820X13496248. PMID 23908302
- [Background] Ong MW, Bashir SJ. Fractional laser resurfacing for acne scars: a review. Br J Dermatol. 2012 Jun;166(6):1160-9. doi: 10.1111/j.1365-2133.2012.10870.x. Epub 2012 May 8. PMID 22296284
- [Background] Manuskiatti W, Triwongwaranat D, Varothai S, Eimpunth S, Wanitphakdeedecha R. Efficacy and safety of a carbon-dioxide ablative fractional resurfacing device for treatment of atrophic acne scars in Asians. J Am Acad Dermatol. 2010 Aug;63(2):274-83. doi: 10.1016/j.jaad.2009.08.051. PMID 20633798
- [Background] Wolfe JW, Butterworth JF. Local anesthetic systemic toxicity: update on mechanisms and treatment. Curr Opin Anaesthesiol. 2011 Oct;24(5):561-6. doi: 10.1097/ACO.0b013e32834a9394. PMID 21841477
- [Background] Hahn IH, Hoffman RS, Nelson LS. EMLA-induced methemoglobinemia and systemic topical anesthetic toxicity. J Emerg Med. 2004 Jan;26(1):85-8. doi: 10.1016/j.jemermed.2003.03.003. PMID 14751483
- [Background] Haedersdal M, Sakamoto FH, Farinelli WA, Doukas AG, Tam J, Anderson RR. Fractional CO(2) laser-assisted drug delivery. Lasers Surg Med. 2010 Feb;42(2):113-22. doi: 10.1002/lsm.20860. PMID 20166154
- [Background] Bachhav YG, Heinrich A, Kalia YN. Controlled intra- and transdermal protein delivery using a minimally invasive Erbium:YAG fractional laser ablation technology. Eur J Pharm Biopharm. 2013 Jun;84(2):355-64. doi: 10.1016/j.ejpb.2012.11.018. Epub 2012 Nov 30. PMID 23207321
- [Background] Haak CS, Farinelli WA, Tam J, Doukas AG, Anderson RR, Haedersdal M. Fractional laser-assisted delivery of methyl aminolevulinate: Impact of laser channel depth and incubation time. Lasers Surg Med. 2012 Dec;44(10):787-95. doi: 10.1002/lsm.22102. Epub 2012 Dec 4. PMID 23212624
- [Background] Haak CS, Bhayana B, Farinelli WA, Anderson RR, Haedersdal M. The impact of treatment density and molecular weight for fractional laser-assisted drug delivery. J Control Release. 2012 Nov 10;163(3):335-41. doi: 10.1016/j.jconrel.2012.09.008. Epub 2012 Sep 21. PMID 23000695
- [Background] Tierney EP, Hanke CW. Fractionated carbon dioxide laser treatment of photoaging: prospective study in 45 patients and review of the literature. Dermatol Surg. 2011 Sep;37(9):1279-90. doi: 10.1111/j.1524-4725.2011.02082.x. PMID 22988990
- [Background] Paasch U, Haedersdal M. Laser systems for ablative fractional resurfacing. Expert Rev Med Devices. 2011 Jan;8(1):67-83. doi: 10.1586/erd.10.74. PMID 21158542
- [Background] Farkas JP, Richardson JA, Burrus CF, Hoopman JE, Brown SA, Kenkel JM. In vivo histopathologic comparison of the acute injury following treatment with five fractional ablative laser devices. Aesthet Surg J. 2010 May-Jun;30(3):457-64. doi: 10.1177/1090820X10373060. PMID 20601578
- [Background] Hantash BM, Bedi VP, Chan KF, Zachary CB. Ex vivo histological characterization of a novel ablative fractional resurfacing device. Lasers Surg Med. 2007 Feb;39(2):87-95. doi: 10.1002/lsm.20405. PMID 17115384
- [Background] Taudorf EH, Haak CS, Erlendsson AM, Philipsen PA, Anderson RR, Paasch U, Haedersdal M. Fractional ablative erbium YAG laser: histological characterization of relationships between laser settings and micropore dimensions. Lasers Surg Med. 2014 Apr;46(4):281-9. doi: 10.1002/lsm.22228. Epub 2014 Feb 5. PMID 24500855